CLINICAL TRIAL: NCT06100835
Title: Enjoy Physical Activity to Battle Sedentary Behaviour and Inactivity Among Older Adults From a Socially Inclusive Perspective (JOIN4JOY).
Brief Title: Feasibility of the JOIN4JOY Programme to Reduce Sedentary Behaviour and Increase Physical Activity in Older Adults.
Acronym: JOIN4JOY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: European Commission (Other); Fundació Blanquerna (Unknown); Fundació Salut i Envelliment (Unknown); Syddansk Universitet (Unknown); Istituto Europeo per lo Sviluppo socio economico Associazione (Unknown); Sport Initiative et Loisir Bleu Association (Unknown); Agaplesion Bethesda Klinik Ulm (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uvicucc_JOIN4JOY
Record Dates: First submitted 2023-09-07; First posted 2023-10-25 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Physical Inactivity; Sedentary Behavior
Keywords: physical activity; joy; social inclusion; older adults; sedentary behaviour; sedentary behavior; nursing homes; enjoyment
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Social Inclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Complex intervention involving physical activity and behaviour change techniques — The intervention protocol derives from a previous, extensive, co-creation phase involving end-users as well as relatives, experts, professionals working working with older adults, university students and researchers.
  It will be based on a structured group-based PA programme supervised by trained professionals, tailored to participants' needs to include joyful components combined with self-management strategies to encourage behaviour change also beyond the sessions. All participants (including end-users but not only) will also be encouraged to join virtual communities of practice (VCoP) for further support and knowledge exchange.

SUMMARY:
Physical activity (PA) and sedentary behavior (SB) programmes for older people in the community and long-term care facilities traditionally focus on achieving functional and health improvements. These approaches face frequent challenges in reaching older people with more social disadvantages and in achieving and maintaining attendance. The aim is to evaluate the acceptability, implementation process and potential impact of a co-created JOIN4JOY PA programme focused on enjoyment and social inclusion for 65+-year-old community-dwelling adults as well as for 65+-year-olds nursing-home residents who live in nursing homes.

DETAILED DESCRIPTION:
Physical activity (PA) and sedentary behavior (SB) programmes for older people in the community and long-term care facilities traditionally focus on achieving functional and health improvements. These approaches face frequent challenges in reaching older people with more social disadvantages and in achieving and maintaining attendance. The aim is to evaluate the acceptability, implementation process and potential impact of a co-created JOIN4JOY PA programme focused on enjoyment and social inclusion for 65+-year-old community-dwelling adults as well as for 65+-year-olds nursing-home residents who live in nursing homes.

Two related multicentric, pragmatic, feasibility studies using mixed methods will be conducted. The programme consists of a novel, co-created PA intervention focusing on enjoyment and social inclusion, grounded in self-management strategies to promote behaviour change. Participants will be offered one weekly, 1-hour session of structured, supervised PA and encouraged to hold more active lifestyles and engage in autonomous physical activity practice. Group sessions will take place in the participant's nursing home or in collaborating social institutions in the community.

Participants will additionally be invited to join virtual communities of practice. At least 72 end-users will be recruited for each setting in 5 European countries (i.e., Spain, Denmark and Italy will focus on the community settings while and Spain, Germany, and France will do so inon nursing homes). The implementation process and its acceptability will be assessed for acceptability, fidelity, participation and satisfaction by means ofwill be assessed by semi-structured interviews, field diaries of sessions and quantitative 5-point Likert-type scales. To evaluate the potential impact, physical function (Short Physical Performance Battery test), quality of life (EUROQOL-5D scale), enjoyment (Physical Activity Enjoyment Scale), perceived improvement (Patient Global Impression of Improvement scale), activities of daily living (Barthel index) and SB patterns (accelerometers) will be assessed. SPSS software will be used for the analysis of quantitative variables with paired t-tests. Qualitative data collected . Ppre- and post-intervention changes will be assessed using determined themathematic analysis following the steps described by of qualitative data.will follow the Braun and Clarke steps.

Ethics and dissemination: A favorable report by the Research Ethics Committee of UVic-UCC (282/2023) was obtained on June 26th, 2023. Participation and withdrawal will be voluntary. When necessary, written permission by the legal guardian will be requested. A broad action of dissemination and communication activities will be targetting both the scientific and the general public.

ELIGIBILITY:
Inclusion criteria for participants in JOIN4JOY-C include:

* Being 65 years of age or above.
* Living in the community.
* No cognitive decline as per short form Mini-Mental State Examination (SMMSE).

Exclusion criteria for participants in JOIN4JOY-C:

* Health condition that contraindicates physical exercise interventions (as per Physical Activity Readiness Questionnaire, PAR-Q).

Inclusion criteria for participants in JOIN4JOY-NH include:

* Being 65 years of age or above.
* Living in a nursing home.
* Ability to participate in group-based, structured PA.

Exclusion criteria for participants in JOIN4JOY-NH include:

* Severe cognitive decline (7 points or above as per Global Deterioration Scale of Reisberg, reported by professional caregivers).
* Severe dependence that requires being bed-bound.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported Physical activity | Before (week 0) and after (week 13)
  measured with de Physical Activity Questionnaire (IPAQ) - Short Form.
Physical activity level | Before (week 0) and after (week 13)
  Measured via Accelerometry . For 7 consecutive days before, and 7 consecutive days after the JOIN4JOY PA programme.
Sedentary Behavior | Before (week 0) and after (Week 13)
  Assessed via the Sedentary Behaviour Questionnaire (SBQ),

SECONDARY OUTCOMES:
Physical function | Before (week 0) and after (week 13)
  Short Physical Performance Battery (SPPB) test,
Quality of life | Before (week 0) and after (week 13)
  EUROQOL-5D-5L scale
Perceived improvement | Before (week 0) and after (week 13)
  Patient Global Impression of Improvement (PGI-I) scale
Enjoyment | After end of physical activity sessions (week 13)
  Physical Activity Enjoyment Scale (PACES)
Sense of community | Before (week 0) and after (week 13)
  Sense of community index (SCI-2)
Participation in the virtual communities of practice | Through study completion and follow-up (estimated 6 months).
  Number of entries in virtual communities of practice, per individual.
Quality of interactions in the virtual communities of practice | Through study completion and follow-up (estimated 6 months).
  Assessed subjectively by the researchers
Degree of satisfaction | Post intervention (week 13)
  5-point Likert Scale
Participation in physical activity sessions | Intervention duration (weeks 1 through 12)
  Field diaries to be completed by trainers on a weekly basis

CONTACTS AND LOCATIONS:
Overall Officials: Laura Coll-Planas, MD, Principal Investigator — University of Vic - Central University of Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coll-Planas L, Fuente-Vidal A, Jerez-Roig J, Karkauskiene E, Romero-Mas M, Intxaurrondo A, Caserotti P, Skjodt M, Dallmeier D, Lefebvre G, Bassinah L, Forgione D, Castro R, Minobes-Molina E, Pares-Martinez C, Blancafort Alias S, Roman-Vinas B, Socorro-Cumplido JL, Nieto-Guisado A, Sansano-Nadal O, Gine-Garriga M. Boosting enjoyment and social inclusion to increase physical activity and reduce sedentary behaviour among older adults: protocol for a feasibility study to test the JOIN4JOY approach in five European countries. BMJ Open. 2024 Jul 27;14(7):e083291. doi: 10.1136/bmjopen-2023-083291. PMID 39067876
- See also: Project official website — https://join4joy.eu/